CLINICAL TRIAL: NCT04929275
Title: Feasability and Impact of Enhanced Recovery Programs After Surgery for Small Bowel Obstruction
Brief Title: Enhanced Recovery Programs and Small Bowel Obstruction
Acronym: RACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A01015-36
Record Dates: First submitted 2021-05-29; First posted 2021-06-18 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2021-05

CONDITIONS: Small Bowel Obstruction; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced recovery program (Other)
  Interventions: Procedure: Enhanced recovery program

INTERVENTIONS:
Procedure: Enhanced recovery program — 12 items of program (preoperative, peroperative postoperative) according to the enhanced recovery after surgery society

SUMMARY:
Small bowel obstruction surgery is frequent and would benefit from enhanced recovery programs. While some studies advocate for their feasibility, it has never been proved and prospective studies are required to confirm the feasibility of such program and the impact on postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adhesionnal small bowel obstruction requiring surgical management

Exclusion Criteria:

* No surgery
* Patients disagreeing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
occurence rate of postoperative ileus | within 30 postoperative days

SECONDARY OUTCOMES:
Feasibility of the enhanced recovery program after small bowel obstruction surgery | within 30 postoperative days
  The feasibility of the enhanced recovery program will be assessed by using the ratio: number of items of the programs followed/ number of items in the programs
Postoperative morbidity | within 30 postoperative days
length of stay | the day of discharge assessed up to 30 days
Rate of nasogastric tube replacement | within 30 postoperative days
Rate of tolerance to solid food | within 30 postoperative days
Time to GI function recovery | within 30 postoperative days
acceptability toward the enhanced recovery program | the day of discharge up to 30 days
  The acceptability will be assessed through 2 qualitative questions and a 1-10 satisfaction scale

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Venara, MD PhD, Principal Investigator — UH Angers
Locations (1):
- UH Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] M L, G B, F F, M B, M D, E PS, Jf H, A V. Enhanced recovery programs following adhesive small bowel obstruction surgery are feasible and reduce the rate of postoperative ileus: a preliminary study. Langenbecks Arch Surg. 2024 Jun 20;409(1):191. doi: 10.1007/s00423-024-03389-7. PMID 38900305